CLINICAL TRIAL: NCT03559413
Title: Prospective Phase I/II Study: Patient-individualized Peptide Vaccination Based on Whole Exome Sequencing With Adjuvant GM-CSF (Granulocyte Macrophage Colony-stimulating Factor) in Children and Young Adults With Primary/Relapsed Acute Lymphoblastic Leukemia
Brief Title: Patient-individualized Peptide Vaccination Based on Tumor-specific Mutations in Children and Young Adults With Primary/Relapsed ALL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Children's Hospital Tuebingen (Other)
Collaborators: German Cancer Research Center (Other); Universität Tübingen (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Peter Lang, Prof. Dr. med., University Children's Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVAC-ALL-1; 2015-005281-29 (EudraCT Number)
Record Dates: First submitted 2018-06-13; First posted 2018-06-18 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Primary/Relapsed Acute Lymphoblastic Leukemia (ALL) of Childhood, Adolescents and Young Adults
Keywords: Individualized peptide vaccination; Immunotherapy; Tumor-specific mutations; Neoantigens
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Biological: Individual peptide vaccination with adjuvant GM-CSF and Imiquimod

INTERVENTIONS:
Biological: Individual peptide vaccination with adjuvant GM-CSF and Imiquimod — Intradermal injection of a cocktail of 3-5 individual HLA-binding peptides. Subcutaneous injection of adjuvant GM-CSF at vaccination site. Topical administration of Imiquimod at vaccination site.

SUMMARY:
The aim of this clinical study is to evaluate the feasibility and safety of an individualized peptide vaccination approach in patients with acute lymphoblastic leukemia (ALL). For this purpose, tumor-specific mutations are analyzed by comparative exome sequencing of tumor and healthy reference tissue. Expression of variants is further validated by RNA sequencing. In a second step, HLA-binding (human leukocyte antigen-binding) peptides derived from mutated protein sequences are selected for vaccination. The peptides are administered as a vaccination cocktail with adjuvant GM-CSF and Imiquimod over a course of 9 months and a total of 16 vaccinations. Primary objective is the de novo induction of a specific T cell response without unacceptable toxicity and acute GvHD (graft versus host disease).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients and young adults with ALL (T, B, pro-B, pre-B or c-ALL) ≥CR3 or with ≥1st relapse after stem cell transplantation (SCT); or patients in ≤CR2 who have received SCT without having reached a sufficient molecular remission prior to, or after SCT (defined as MRD ≥10^-4); or patients with initially refractory disease to standard treatment who could proceed to stem cell transplantation with alternative treatment options.
* Hematological remission has to be reached (<5% blasts in bone marrow or detectable minimal residual disease (MRD) ≤5x10^-2) after salvage chemotherapy and/or subsequent SCT.

Exclusion Criteria:

* Frank relapse (>5% leukemic blasts).
* Ejection fraction <25%; Creatinine-clearance <40ml/min; Bilirubin >4mg/dl, Transaminases >400 units/ml; severe infection (HIV, Hepatitis), acute GvHD III-IV or chronic GvHD.
* Significant psychiatric disabilities, uncontrolled seizure disorders or severe peripheral neuropathy/ leukoencephalopathy.
* Signs of autoimmune disease (i.e. idiopathic thrombocytopenic purpura, autoimmune hemolytic anemia).
* Need for immunosuppressive drugs.
* No tumor material available for exome sequencing.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is "success of treatment" defined as a patient showing a vaccination-induced T-cell response without unacceptable toxicity and acute GvHD of Grade III or higher or extensive chronic GvHD until day 120 (after 10 vaccinations). | 120 days
  Side effects wil be assessed according to NCI common toxicity criteria V4.0. GvHD will be graded according to Glucksberg criteria. A vaccine-specific response will be defined by an at least 2-fold elevated cytokine expression of CD4+ and/or CD8+ T cells over background in response to stimulation with the vaccine peptides. A vaccine-induced response will be defined by an at least 2-fold elevated response at a certain timepoint compared to pre-vaccination.

SECONDARY OUTCOMES:
To evaluate CD4+ and/or CD8+ T-cell responses over the vaccination period. | 246 days
  T-cell responses will be measured after completion of the study at day 246 and will be analyzed with regard to the T-cell responses at day 120.
To evaluate changes in minimal residual disease (MRD) during and after treatment. | 246 days
  Possible reduction of MRD levels on days 36, 120 and 246 (after 7, 10 and 16 vaccinations) measured as reduction of 1 log compared to baseline yes/no.
To evaluate the relapse rate during and after treatment. | 246 days
  Relapse rates will be assessed on days 120 and 246.
To evaluate the event-free survival (EFS) during and after treatment. | 246 days
  EFS will be assessed on days 120 and 246.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lang, Prof. Dr., Principal Investigator — University Children's Hospital Tuebingen
Locations (5):
- Germany (5):
  - University Medical Center for Children and Adolescents Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Children's Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - University Children's Hospital Munich, Center for Pediatric Hematology and Oncology, München, Bavaria
  - University Hospital Düsseldorf, Clinic for Pediatric Oncology, Hematology and Clinical Immunology, Düsseldorf, North Rhine-Westphalia
  - Charite Universitätsmedizin Berlin, Department of Pediatric Oncology/Hematology, Berlin

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting at time of publication
Access Criteria: Anyone, upon request to PI